CLINICAL TRIAL: NCT05169125
Title: Effect of Reducing Dialysate Sodium Concentration on Blood Pressure Variability in Hemodialysis Patients: A Randomized Controlled Trial
Brief Title: Reducing Dialysate Sodium Effect on Blood Pressure Variability in Hemodialysis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Hadeer Tarek Abdelaziz Gomaa, principal investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MS.21.06.1547
Record Dates: First submitted 2021-11-10; First posted 2021-12-23 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: Hemodialysis Patients
Keywords: sodium; variability; hemodialysis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: standard hemodialysis. (Active Comparator): patients who will undergo standard hemodialysis (dialysate sodium concentration 143 mmoL/L)
  Interventions: Procedure: standard hemodialysis
- Group B: lower dialysate sodium hemodialysis. (Active Comparator): patients who will undergo hemodialysis with lower dialysate sodium concentration (140 mmoL/L).
  Interventions: Procedure: lower dialysate sodium dialysis

INTERVENTIONS:
Procedure: standard hemodialysis — patients who will undergo standard hemodialysis (dialysate sodium concentration 143 mmoL/L)
  Arms: Group A: standard hemodialysis.
Procedure: lower dialysate sodium dialysis — patients who will undergo hemodialysis with lower dialysate sodium concentration (140 mmoL/L)
  Arms: Group B: lower dialysate sodium hemodialysis.

SUMMARY:
In this study the investigators aim to test the effect of lowering dialysate sodium concentration on visit-to-visit blood pressure variability in hemodialysis patients who have achieved their dry weight.

DETAILED DESCRIPTION:
Cardiovascular diseases are considered the major cause of mortality in maintenance hemodialysis patients. Nevertheless, hypertension is recognized as an important modifiable risk factor for cardiovascular disease among hemodialysis (HD) patients.

Apart from blood pressure levels, BP variability, which reflects the fluctuation in BP, has been described as an independent risk factor that linearly associated with all-cause and cardiovascular mortality in HD patients.

BPV is categorized as either long or short term, based on the time interval over which it is considered. In the dialysis population, long-term BPV is typically defined on the basis of BP measurements taken at the start of each thrice-weekly hemodialysis treatment (interdialytic BPV). On the other hand, short-term BPV among dialysis patients can be considered in terms of variability that occurs during hemodialysis treatments (intradialytic BPV). Researchers believed that the mitigation strategies of BPV must be paid attention to.

Sodium load is associated with thirst, fluid retention, interdialysis weight gain and hypertension for hemodialysis patients, therefore the Kidney Disease Outcomes Quality Initiative (KDOQI) Clinical Practice Guideline highlighted the importance of limiting sodium intake and adequate sodium removal which is considered one of the most important goals of the dialysis therapy.

Interestingly, a recent study showed that mild decrease in dialysate sodium concentration could improve systolic blood pressure variability in HD patients at their dry weight, thus improving blood pressure complications and subsequent complications. However, whether improving sodium balance could potentially contribute to better BPV management in HD patients has not been assessed in a randomized manner. Therefore, this study aims to investigate whether lowering dialysate sodium concentration could help mitigate long term (interdialytic) BPV in hemodialysis patients in a randomized controlled manner.

ELIGIBILITY:
Inclusion Criteria:

* Patients' age ≥18 years
* Patients who had been on regular hemodialysis for at least 3 months.
* Patients' residual daily urine output is less than 100 mL/day.
* Pre study one week average systolic BP ≥120 mmHg but ≤ 180 mmHg.
* Patients who have achieved their dry weight as assessed by clinical examination.
* Predialytic serum sodium level ≥ 140mmol/l.
* Kt/V ≥ 1.2

Exclusion Criteria:

* Patients who have advanced heart failure or permanent atrial fibrillation decompensated liver disease, neoplastic illness, overt edema.
* History of acute cardiovascular accidents or infections during 3 months preceding entry into the study.
* Patients prone to hypotension or other intradialytic adverse events.
* Patients participating in another interventional study that may affect blood pressure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
blood pressure variability. | 2 weeks after the study duration (3 months).
  visit to visit blood pressure variability in both groups.

SECONDARY OUTCOMES:
interdialytic weight gain | 2 weeks after the study duration (3 months).
  interdialytic weight gain
antihypertensive medication regimen | 2 weeks after the study duration (3 months).
  antihypertensive medication regimen
the frequency of intradialytic adverse events | 2 weeks after the study duration (3 months).
  the frequency of intradialytic adverse events as hypotensive crises and cramps.

CONTACTS AND LOCATIONS:
Overall Officials: Ghada El-said, Ass. Prof., Study Chair — Mansoura University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abdulaziz HMM, Gomaa H, El-Said G. Improvement of visit-to-visit SBP variability with lowering dialysate sodium concentration in patients undergoing hemodialysis: a randomized controlled trial. J Hypertens. 2026 Jan 23. doi: 10.1097/HJH.0000000000004243. Online ahead of print. PMID 41649081
- [Derived] Marshall MR, Wang MY, Vandal AC, Dunlop JL. Low dialysate sodium levels for chronic haemodialysis. Cochrane Database Syst Rev. 2024 Nov 5;11(11):CD011204. doi: 10.1002/14651858.CD011204.pub3. PMID 39498822